CLINICAL TRIAL: NCT07001332
Title: ELEVATE High-Risk PCI Pivotal Study
Acronym: ELEVATE III
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magenta Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRD-0001723
Record Dates: First submitted 2025-05-07; First posted 2025-06-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: High-Risk Percutaneous Coronary Intervention (High-risk PCI)

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, open-label, interventional, randomized, and controlled study with an active control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Elevate (Experimental): Subjects receiving the Elevate System
  Interventions: Device: Elevate
- Impella (Active Comparator): Subjects receiving the Impella System
  Interventions: Device: Impella

INTERVENTIONS:
Device: Elevate — The Elevate System is a catheter- mounted, self-expanding and retrievable, continuous-flow pump, designed to unload the left ventricle by actively transporting blood from the left ventricle into the ascending aorta, thus augmenting cardiac output and maintaining systemic arterial pressure during complex/high-risk coronary interventions. Subjects will receive an Elevate prior to their high-risk percutaneous intervention.
  Arms: Elevate
Device: Impella — Subjects will receive an Impella prior to their high-risk percutaneous intervention.
  Arms: Impella

SUMMARY:
The ELEVATE III Pivotal Study is a prospective, multi-center, open-label, interventional, randomized, controlled study with an active control group. The study is intended to assess the safety and efficacy of the Elevate™ percutaneous Left Ventricular Assist Device System in patients referred to high-risk percutaneous coronary interventions (HR-PCI).

DETAILED DESCRIPTION:
The Elevate™ percutaneous Left Ventricular Assist Device System is a temporary (≤ 6 hours) ventricular support device indicated for use during high-risk percutaneous coronary interventions (HR-PCI) performed electively or urgently in hemodynamically stable patients with severe coronary artery disease. Use of the Elevate™ System in these patients may prevent hemodynamic instability, which can result from repeat episodes of reversible myocardial ischemia that occur during planned temporary coronary occlusions.

ELIGIBILITY:
Inclusion Criteria:

1. Non-emergent, percutaneous coronary intervention is planned on at least one stenotic lesion of a native coronary artery or bypass graft (de novo or restenosis).
2. A heart team that includes an interventional cardiologist and cardiac surgeon has determined that HR- PCI is an appropriate therapeutic option.
3. Participant signed the informed consent.

Exclusion Criteria:

1. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure.
2. Prior stroke with any permanent, significant (mRS>2) neurological deficit, or stroke or TIA within 3 months prior to enrollment.
3. Any condition or scheduled surgery that will require discontinuation of the antiplatelet and/or anticoagulation therapy within 90 days of the index procedure.
4. Evidence of left ventricular thrombus.
5. Aortic valve stenosis/calcification (valve area ≤ 1.5 cm2).
6. ≥ Moderate aortic valve regurgitation (≥ 2+ on a 4-grade scale by transthoracic echocardiography).
7. Femoral access site incompatibility that precludes placement of either the Treatment or Control device.
8. Patient on dialysis.
9. Known or suspected coagulopathy OR abnormal coagulation parameters.
10. Known allergy, sensitivity or intolerance to nickel.
11. Infection of the proposed procedural access site; OR suspected systemic active infection, including any fever or known active COVID-19 infection.
12. Allergy, sensitivity or intolerance to heparin, or contrast media, including known heparin-induced thrombocytopenia (HIT).
13. Any non-cardiac condition with a life expectancy < 12 months.
14. Subject participation in another investigational drug or device trial (with the exception of post-market registries and observational studies, subject to Sponsor review and approval).
15. Pregnancy or breast-feeding.
16. Subject has other medical, social, or psychological problems that, in the opinion of the Investigator, compromise the participant's ability to provide written informed consent and/or to comply with study procedures.
17. Subject belongs to a vulnerable population.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
A composite of the incidence of major safety and effectiveness parameters. | 30 days
  A composite of the incidence of: 1. Major Adverse Cardiac and Cerebrovascular Events (MACCE): Death, Myocardial Infarction, Stroke or Transient Ischemic Attack, Unplanned Repeat Revascularization; 2. Major intra-procedural hemodynamic events on Mechanical Circulatory Support: Severe Hypotension, Cardio-Pulmonary Resuscitation or Cardioversion; 3. Major Mechanical Circulatory Support-related access site complications: Vascular Injury Requiring Intervention or Access Site Bleeding.

SECONDARY OUTCOMES:
Major Hemolysis during index hospitalization | Perioperative/Periprocedural
  Incidence of Major Hemolysis
Incidence of Bleeding Academic Research Consortium (BARC) Type 3 or Type 5 bleeding events related to the index percutaneous coronary intervention. | Perioperative/Periprocedural
  The incidence of bleeding events related to the index percutaneous coronary intervention meeting the definition of Bleeding Academic Research Consortium (BARC) Type 3 or Type 5 bleeding.
Length of hospital stay | Perioperative/Periprocedural
  Length of hospital stay across all enrolled patients
Length of ICU/CCU stay | Perioperative/Periprocedural
  Length of ICU/CCU stay across all enrolled patients

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Tampa General/USF, Tampa, Florida
  - Wellstar Health System, Marietta, Georgia
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Maimonides Health, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone/Bellevue/Long Island, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Advocate Aurora Health Research Institute- St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No